CLINICAL TRIAL: NCT06065592
Title: Unveiling Prognosis Cancer-Associated Thromboembolism Biomarkers and Their Related Polymorphisms: Exploring Their Involvement With Immune Circulating Cells and Therapeutic Reversibility
Brief Title: Exploring Cancer-Associated Thromboembolism Prognosis Biomarkers and Polymorphisms
Acronym: CAT_PB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese University (Other)
Collaborators: Haykel Hospital (Unknown)
Responsible Party: Principal Investigator, Nehman Makdissy, Principal Investigator, Professor, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lebanese University
Record Dates: First submitted 2023-09-06; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Solid Tumor; Thromboembolism; Cardiovascular Diseases; Immune System Diseases; Inflammatory Diseases; Colon Cancer; Breast Cancer; Prostate Cancer; Hepatocellular Carcinoma; Lung Cancer; Chemotherapy; Immunotherapy
Keywords: cancer; thromboembolism; cardiovascular; immune cells; immunotherapy; chemotherapy; inflammation; gene polymorphism; biomarker; LncRNA; Palbociclib; Rivaroxaban; blood coagulation
MeSH Terms: conditions — Neoplasms; Thromboembolism; Cardiovascular Diseases; Immune System Diseases; Colonic Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Inflammation; Thrombosis | interventions — palbociclib; Rivaroxaban

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Non-Carriers of Targeted Gene-Related Polymorphisms (GRPs) in Cancer Patients (Active Comparator): Cancer patients without any incidence of thromboembolism will be included if they are non-carriers of the targeted gene-related polymorphism (GRP).
  Interventions: Genetic: SNP
- Carriers of Targeted GRPs in Cancer Patients (Active Comparator): Cancer patients without any incidence of thromboembolism will be included if they are carriers of the targeted gene-related polymorphism.
  Interventions: Genetic: SNP
- Carriers of Targeted GRPs in Cancer-Associated Thromboembolism Patients (Experimental): Cancer patients with incidence of thromboembolism will be included if they are carriers of the targeted gene-related polymorphism.
  Interventions: Genetic: SNP
- Carriers of Targeted GRPs in Cancer-Associated Thromboembolism Patients Treated with Palbociclib (Experimental): Cancer patients with incidence of thromboembolism will be included if they are carriers of the targeted gene-related polymorphism and will be subjected to Palbociclib treatment.
  Interventions: Drug: Palbociclib; Genetic: SNP
- Carriers of Targeted GRPs in Cancer-Associated Thromboembolism Treated with Anti-Coagulant (Experimental): Cancer patients with incidence of thromboembolism will be included if they are carriers of the targeted gene-related polymorphism and will be subjected to anti-coagulant treatment.
  Interventions: Drug: Rivaroxaban; Genetic: SNP

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered at a dose of 125 mg oral on a 21/7 cycle.
  Other Names: Ibrance
  Arms: Carriers of Targeted GRPs in Cancer-Associated Thromboembolism Patients Treated with Palbociclib
Drug: Rivaroxaban — Rivaroxaban will be administered at a dosage of 15 mg intravenously twice a day for 21 days, followed by 20 mg once daily for the subsequent 21 days.
  Other Names: Xarelto
  Arms: Carriers of Targeted GRPs in Cancer-Associated Thromboembolism Treated with Anti-Coagulant
Genetic: SNP — diagnostics of patients' carriers or not of the risk allele(s)
  Other Names: Risk Allele(s)

SUMMARY:
This study aims to assess biomarkers and their related polymorphisms in the context of cancer-associated thromboembolism, with a particular focus on their interaction with the immune system. The roles of immune checkpoints, inflammatory and angiogenesis factors, as well as circulating immune cells will be elucidated. Additionally, our investigation extends to the exploration of long non-coding RNAs (LncRNAs) and genes associated with the coagulation vascular system. Initially, these aspects will be evaluated in the context of colorectal cancer, with the intention to expand our research to other solid tumors.

The identification of these biomarkers and genetic factors holds the potential to revolutionize therapeutic approaches for patients with cancer-associated thromboembolism, shedding light on their chemotherapy resistance. The effectiveness of combining immunotherapy with targeted inhibitors like Palbociclib and anticoagulants such as Rivaroxaban, among other potential interventions, will be assessed.

This study aims to make significant contributions to the understanding of these critical aspects, ultimately leading to the development of more effective treatment strategies for cancer patients.

DETAILED DESCRIPTION:
Cancer, especially solid tumors, remains a significant global health challenge despite ongoing advancements in risk factor identification and targeted therapies. Among the various complexities of cancer treatment, the relationship between cancer and thromboembolism, characterized by arterial and venous thrombosis, has attracted attention due to its significant impact on patient outcomes.

Cancer cells activate the coagulation system, leading to prothrombotic disorders in the vascular wall and promoting tumor progression. Patients with cancer, particularly those undergoing systemic chemotherapy, face an increased risk of thromboembolism due to abnormal blood clotting mechanisms.

Recent research has emphasized the importance of identifying novel biomarkers for risk assessment, prognosis determination, and treatment selection in cancer. Among these biomarkers, long non-coding RNAs (LncRNAs) and those of the vascular coagulation system have emerged as pivotal players in cancer development and progression. However, their role as prognostic and predictive biomarkers for cancer risk and treatment response remains relatively unexplored.

Understanding the complex interplay between cancer, immune responses, and thromboembolism is crucial. Immunological subsets, including central immune effector T cells (CD8+, CD25+), NK cells, and macrophages, have been linked to cancer prognosis. Furthermore, therapies that modulate the immune system, such as immunotherapy and cell-based therapies, hold promise for improving cancer treatment outcomes.

Most notably, these therapies exhibit immunomodulatory effects, triggering immunogenic cell death and preventing immunosuppression. However, their efficacy may be compromised in cases of cancer associated with clotting abnormalities within the circulatory system. Progenitor cells, including stem cells and endothelial progenitor cells (EPCs), are emerging as potential players in cancer therapy, offering new avenues for research.

Among the innovative approaches is the assessment of circulating immune and endothelial progenitor cells (termed "CIEs"), which may play significant roles in the mechanisms underlying cancer-associated thromboembolism. Understanding the relationship between these cells, inflammatory and angiogenic factors, immune checkpoint, and cancer progression could pave the way for improved cancer risk assessment and treatment strategies.

This study seeks to contribute to our understanding of the intricate connections between LncRNA, coagulation-related biomarkers, thromboembolism, immune responses, and cancer, using solid tumors as a representative example. By shedding light on these complex interactions, this study aims to identify potential biomarkers that can guide risk assessment and treatment decisions, ultimately improving the management of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of white ethnicity.
* Age between > 18
* Both males and females.
* Diagnosis of selected cancer type (e.g., colorectal cancer).
* Cancer stage 0/I/II without metastasis or lymph node dissemination at the time of enrollment.
* No previous cancer therapy (radiotherapy, chemotherapy, or immunotherapy) received before study enrollment.
* Unrelated patients.

Exclusion Criteria:

* Cancer stage III/IV.
* History of hematological cancer types or previous cancers, recurrent or relapse.
* Diagnosis of inflammatory bowel diseases.
* Pre-existing cardiovascular diseases or coronary artery diseases.
* Confirmed treated or untreated autoimmune diseases.
* Metabolic disorders, diabetes, or hypertension.
* Neurological diseases.
* Evidence of cardiac, renal, bone, or cerebral damage.
* Presence of more than one type of malignancies.
* Active infections or myositis.
* Familial polyposis.
* Alcohol or smoking habits.
* Colon-affecting food allergies.
* Body mass index (BMI) >30.
* Significant weight loss within the last 2 years.
* History of abdominal surgeries.
* Pregnancy.
* Related patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Venous Thromboembolism (VTE) Events including: Deep Vein Thrombosis (DVT), Pulmonary Embolism (PE), and other Thromboembolic Events (Vein Thrombosis, Portal Vein Thrombosis, Superior Mesenteric Vein Thrombosis, and Renal Vein Thrombosis) | up to 60 months
  The outcome measure of VTE including DVT, PE, and other thromboembolic events will be assessed by : (1) Clinical Assessment: Clinical symptoms such as swelling and pain in the lower limbs, tenderness behind the lower leg and/or medial thigh, and supplementary evaluation with color ultrasound of the veins in both lower limbs (lower extremity venography); (2) Imaging: CT pulmonary arteriography (CTPA) will be employed in conjunction with related clinical manifestations such as dyspnea and shortness of breath for diagnosing PE; (3) Laboratory Criteria: Diagnostic criteria will also consider laboratory parameters, including elevated D-dimer levels (> 1000 ng/mL), increased fibrinogen levels (> 700 mg/dL), and shortened activated partial thromboplastin time (aPTT) (< 20 sec).
Assessment of Cancer Progression | up to 60 months
  The assessment of cancer progression will be conducted using the standardized TNM staging system and applying the Response Evaluation Criteria (RECIST) guideline (ver. 1.1). Clinical parameters, laboratory tests indicative of cancer progression (including tumor markers and histopathological analysis), and relevant imaging modalities (e.g., CT, MRI, or PET scans) will be employed to evaluate the extent of primary tumor growth, lymph node involvement, and the presence of distant metastases. Progression-Free Survival (PFS), a key primary clinical endpoint for assessing cancer progression, will be calculated as the duration (in months) from the date of enrollment in the study until the tumor progresses, new lesions appear, or until the participant's death from any cause. Cancer progression will be determined based on RECIST guidelines, considering an increase in tumor size or the appearance of new lesions according to imaging assessments and clinical evaluations.
Identification of Potential Biomarkers | Once at the moment of the patient's enrollment in the study
  The objective of this outcome is to identify and characterize novel biomarkers associated with thromboembolism and cancer progression. Specifically, the assessment will focus on Long Non-Coding RNAs (LncRNAs) such as CDKN2B and CDKN2B-AS1, and markers related to the vascular coagulation system including ACE, PAI-1, FXIII, and Prothrombin. This identification process will involve collecting biological samples (e.g., blood, tissue) from enrolled patients at the time of study enrollment. The assessment will analyze and evaluate the expression and polymorphisms of the studied genes (CDKN2B, CDKN2B-AS1, ACE, PAI-1, FXIII, and Prothrombin) using quantitative PCR (qPCR), with Ct (Cycle threshold) as the common unit of measure for all genes. This comprehensive assessment aims to enhance our understanding of the molecular signatures linked to thromboembolism and cancer progression, illuminating potential diagnostic and therapeutic avenues for improved patient outcomes.
Evaluation of Treatment Response to Palbociclib | up to 60 months
  This primary outcome assesses treatment response in patients undergoing Palbociclib therapy for controlling cancer progression and thromboembolism. The evaluation will employ RECIST criteria to measure the percentage change in tumor size, indicative of treatment effectiveness.

SECONDARY OUTCOMES:
Survival Rates | up to 60 months
  Analysis of overall survival and progression-free survival rates among groups
Examination of Genetic Variants, specifically rs1333049 G>C Polymorphism within the CDKN2B-AS1 Gene | Once at the moment of the patient's enrollment in the study
  The objective of this secondary outcome is to examine genetic variants, with a specific focus on the rs1333049 G>C polymorphism within the CDKN2B-AS1 gene. The screening for polymorphism(s) will be determined by genotyping analysis using TaqMan PCR-based genotyping for SNP identification.
Adverse Events | up to 60 months
  Monitoring and reporting of adverse events related to the Palbociclib and Rivaroxaban treatment regimen.
Immunophenotyping of Immune Cell Populations | up to 60 months
  This outcome aims to comprehensively assess immune cell populations involved in the immune response, including T cells, B cells, natural killer (NK) cells, dendritic cells (DCs), and macrophages. The objective is to characterize changes in immune cell subsets over time, providing insights into the immune response dynamics. The assessment will involve immunophenotyping using flow cytometry to quantify and analyze the different immune cell populations. The unit of measure for this assessment will be the percentage of change of T cells, B cells, NK cells, DCs, and macrophages in the total population. The percentage of change will be determined up to a period of 60 months relatively to their levels at the diagnostic time.
Inflammatory Cytokine Profiling | up to 60 months
  This outcome focuses on assessing the levels of cytokines secreted by immune cells, including interferons (IFNs), interleukins (ILs), and tumor necrosis factor (TNF). The objective is to understand cytokine dynamics and their role in the immune response. The assessment will involve cytokine profiling by flow cytometry or ELISA. The levels of IFNs, ILs, and TNF will be measured as a percentage of change over a period of 60 months, relative to their levels at the diagnostic time. This standardized approach of using a common unit of measure will enable a comprehensive and unified evaluation of cytokine variations, providing critical insights into the immune response dynamics throughout the study duration.
Evaluation of Tumor-Infiltrating Lymphocytes (TILs) | up to 60 months
  This outcome aims to evaluate the presence and distribution of TILs within the tumor microenvironment. The objective is to understand the role of TILs in the immune response against the tumor. The assessment will involve analyzing tissue samples for TIL presence and distribution by immunohistochemistry (IHC) or flow cytometry.
Assessment of Immune Checkpoint Expression (e.g., PD-1 and CTLA-4) | up to 60 months
  This outcome focuses on investigating the expression of immune checkpoint molecules, specifically programmed cell death protein 1 (PD-1) and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4). The objective is to understand the role of immune checkpoints in regulating the immune response. The assessment will involve evaluating immune checkpoint expression using techniques such as flow cytometry or PCR. The levels of PD-1 and CTLA-4 expression will be measured in the percentage of change over a period of 60 months, relative to their levels at the diagnostic time. Utilizing a standardized common unit of measure ensures a uniform assessment, allowing for a comprehensive understanding of the immune checkpoint dynamics and their impact on the immune response throughout the study's duration.
Measurement of Angiogenic Factors (e.g., VEGF) | up to 60 months
  This outcome aims to assess alterations in angiogenic factors, with a specific focus on Vascular Endothelial Growth Factor (VEGF), in relation to treatment and study outcomes. VEGF is a key regulator of angiogenesis and is associated with tumor vascularization. The serum concentrations of VEGF-A/C will be measured by ELISA, providing valuable insights into the angiogenic processes linked to the immune response and their potential impact on treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nehman Makdissy, Professor, Study Chair — Lebanese University
Locations (2):
- Lebanon (2):
  - Haykel Hospital, Tripoli, North Lebanon
  - Lebanese University, Tripoli, North Lebanon

IPD SHARING:
Plan to Share IPD: No